CLINICAL TRIAL: NCT03685721
Title: Genotype -Phenotype Correlation of PKLR Variants With Pyruvate Kinase, 2,3-Diphosphglycerate and ATP Activities in Red Blood Cells of Patients With Sickle Cell Disease
Brief Title: Genotype -Phenotype Correlation of PKLR Variants With Pyruvate Kinase, 2,3-Diphosphglycerate and Adenosine Triphosphate Activities in Red Blood Cells of People With Sickle Cell Disease
Status: Recruiting | Type: Observational
Sponsor: National Heart, Lung, and Blood Institute (NHLBI) (NIH)
Responsible Party: Sponsor
Organization: National Institutes of Health Clinical Center (CC) (NIH)
Other Study IDs: 180146; 18-H-0146
Record Dates: First submitted 2018-09-25; First posted 2018-09-26 (Actual); Last update posted 2025-10-14 (Actual); Status verified 2025-09-24

CONDITIONS: Sickle Cell; PKLR Variants; Adenosine Triphosphate Activities
Keywords: ATP; Trait; GDP; Genetics; Natural History

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Cross-Sectional
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (3):
- HbAS: HbAS genotype, of African American descent;Between 18 and 80 years of age
- Healthy control: African American descent;Between 18 and 80 years of age
- SCD: HbSS, HbSC, HbSbeta-thal has sickle cell disease and is of African American descent;Between 18 and 80 years of age

SUMMARY:
Background:

Some people with the same disorder on a genetic level have more complications than others. Researchers want to look for a link between the PKLR gene and sickle cell disease (SCD) symptoms. The PKLR gene helps create a protein, called pyruvate kinase that is essential in normal functioning of the red blood cell. Differences in the PKLR gene, called genetic variants, may cause some changes in the pyruvate kinase protein and other proteins, that can affect functioning of the red blood cell adding to the effect of SCD. Researchers can study these differences by looking at DNA (the material that determines inherited characteristics).

Objective:

To study how the PKLR gene affects sickle cell disease.

Eligibility:

Adults ages 18-80 of African descent. They may have sickle cell disease or not. They must not have had a transfusion recently or have a known deficiency of pyruvate kinase. They cannot be pregnant.

Design:

Participants will be screened with questions.

Participants will have blood drawn by needle in an arm vein. The blood will be genetically tested. Not much is known about how genes affect SCD, so the test results will not be shared with participants or their doctors.

...

DETAILED DESCRIPTION:
Polymerization of deoxy-sickle-hemoglobin (deoxy-HbS), the root cause of sickle cell disease (SCD) is influenced by a few factors, a key factor is 2,3-diphosphoglycerate (2,3-DPG) concentration in the red blood cells. 2,3-DPG is an allosteric effector on hemoglobin oxygen binding with a greater binding affinity to deoxygenated hemoglobin than to oxygenated hemoglobin, thus favoring polymerization of deoxy-HbS. In addition, increased 2,3-DPG concentration decreases intracellular pH in red blood cells which further promotes HbS polymerization.

2,3-DPG is an intermediate substrate in the glycolytic pathway, the only source of ATP production in red blood cells. Pyruvate kinase (PK) is a key enzyme in the final step of glycolysis; PK converts phosphoenolpyruvate (PEP) to pyruvate, creating 50% of the total red cell adenosine triphosphate (ATP) that is essential for maintaining integrity of the red cell membrane. Indeed, PK deficiency (PKD) caused by mutations in the PKLR gene that encodes red cell PK, leads to chronic hemolytic anemia. Reduced PK activity leads to accumulation of the upstream enzyme substrates, including 2,3-DPG. While increased 2,3-DPG concentration and reduction of hemoglobin oxygen affinity is beneficial in anemia caused by PKD, increased 2,3-DPG levels combined with decreased intracellular red cell pH can be detrimental in the presence of HbS, as it favors deoxy-HbS polymerisation, and thereby intravascular sickling. Indeed, the combination of PK deficiency and sickle cell trait causing an acute sickling syndrome has been previously reported in two cases.

PKLR mutations, however, are rare but intraerythrocytic PK enzyme levels form a spectrum which suggest that PKLR is likely to be a quantitative trait gene. A genetic diversity in PKLR with a range of SNPs, including several loss-of-function variants have been described in malaria-endemic populations, some of which have been associated with a significant reduction in attacks with Plasmodium falciparum malaria. These observations suggest that similar to HbS, malaria has led to positive selection of PKLR variants in the same geographic regions.

This study seeks to determine the PKLR genetic diversity in our sickle cell cohort, and whether PKLR variants modify PK levels, and activities of 2,3-DPG and ATP, key players in the sickle pathology. If so, PKLR could be another genetic determinant of SCD severity and phenotype; and increasing PK-R activity, which leads to a decrease in intracellular 2,3-DPG concentration, presents an attractive therapeutic target for SCD.

Several approaches have been considered for targeting the polymerization of deoxy-HbS, the root cause of SCD. In addition to agents inducing fetal hemoglobin, other agents that target HbS polymerization through increasing affinity of hemoglobin for oxygen (eg. GBT440), are in clinical trials (NCT03036813; NCT02850406). The results of this study could form the basis for a clinical trial of AG348, an allosteric activator of PK that is already in clinical Phase 2/3 studies for PK deficiency (NCT02476916), for treating acute sickle cell pain.

ELIGIBILITY:
* INCLUSUION CRITERIA:
* Between 18 and 80 years of age
* African or of African descent

EXCLUSION CRITERIA:

* Self-reported history of blood transfusion within the last 8 weeks
* Known to have pyruvate kinase deficiency and be on AG348
* All volunteers will undergo the consent process under this protocol to allow for eligibility assessment. Once they have been consented to participate, they will undergo procedures per Protocol.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: The study will be listed on the clinicaltrials.gov, Clinical Center research studies, and the National Heart, Lung and Blood Institute patient recruitment websites. Patients who are followed on other NHLBI sickle cell protocols may be asked to participate in this study, particularly subjects enrolled in the Natural History of Sickle Cell Disease (NCT00081523; 04-H-0161).
Sampling Method: Non-Probability Sample
Enrollment: 800 (Estimated)
Dates: Start 2018-10-11 (Actual); Primary Completion 2026-07-01 (Estimated); Study Completion 2026-07-01 (Estimated)

PRIMARY OUTCOMES:
Genotype the 4 PKLR intron-2 variants | Upon enrollment of each subject
  To have genotyped the 4 PKLR intron-2 variants in SCD patients from the NHLBI cohort using genomic DNA and compare them to a cohort of healthy ethnic-matched non-SCD controls and a cohort of sickle cell trait carriers, with those reported in 1000 genome project (http://www.1000genomes.org).
Analysis of PK-R transcriptome in red blood cells | Interim analysis performed for each group N=125
  Have a correlated profile of the PK-R RNA sequence with the 4 PKLR intronic genetic variants.
Correlation of 2,3-DPG, ATP and pyruvate kinase activities with PKLR intron-2 variants | Interim analysis performed for each group N=125
  Assess correlation between the quantitative assays and genotype

CONTACTS AND LOCATIONS:
Overall Officials: Swee Lay Thein, M.D., Principal Investigator — National Heart, Lung, and Blood Institute (NHLBI)
Locations (1):
- National Institutes of Health Clinical Center, Bethesda, Maryland, United States

REFERENCES:
- See also: NIH Clinical Center Detailed Web Page — https://clinicalstudies.info.nih.gov/cgi/detail.cgi?A_2018-H-0146.html